CLINICAL TRIAL: NCT07186712
Title: The Incidence of Early Trauma Induced Coagulopathy and Hyperfibrinolysis in Severely Injured Trauma Patients in the Emergency Room: a Retrospective Cohort Study
Acronym: eTIC
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 1150/2025
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Early Trauma Induced Coagulopathy; Tic
Keywords: eTIC; coagulopathy; trauma
MeSH Terms: conditions — Tics; Hemostatic Disorders; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients in the trauma resuscitation bay of the Medical University of Graz: Valid thrombelastogramm available

SUMMARY:
The aim of this study is to quantify the incidence of eTIC (defined as an elevated appt) and hyperfibrinolysis (defined as Ly30>7) in early trauma patients. To identify patients at risk of eTIC and hyperfibrinolysis, we will conduct a systematic search for trauma patients with an ISS>16 in whom a thrombelastogram (TEG) was obtained in the emergency department (ED)

DETAILED DESCRIPTION:
Despite excessive efforts to reduce the number of preventable deaths in patients suffering from traumatic injuries, hemorrhage is still a leading cause of morbidity and mortality in this patient group. (1) The importance of trauma induced coagulopathy (TIC) on the extent of blood loss has been known at least since 1982. Where Kashuk et al. described the lethal triad of hypothermia, acidosis and coagulopathy for trauma patients. (2) In 2003 two landmark studies firstly identified that coagulopathy was present in the early phase after patients suffered severe traumatic injuries and prior to resuscitation efforts. In both studies the rate of early trauma induced coagulopathy (eTIC) was high (24.4% Brohi et al., 28% Macleod et al.), even in patients with relatively low median injury severity scores (mean ISS 20 and 9). Notably, both studies identified eTIC as an independent predictor of mortality. (3) (4) Nowadays, health care providers and guidelines heavily emphasis the importance of eTIC in trauma resuscitation. However, in a cohort study from Teeter et al. published in 2024 with the data of two major trauma centers in the US found that the incidence of eTIC (defined as the initial prothrombin time (PT) or partial thromboplastin time (PTT) above normal per each center's reference range) increased to 33.4% and that coagulopathy had a major impact on mortality over all severity ranges. (5) However, to detect trauma induced coagulopathy new technologies such as thrombelastography (TEG) and rotational thromboelastometry (ROTEM) have been implemented in the trauma algorithm of major trauma centers since 2003. These tests offer a rapid, comprehensive assessment of the dynamic and sequential processes involved in trauma-induced coagulopathy. (6) With the opportunity of early detection of different entities of eTIC including Hyperfibrinolysis, Thromelastography has shown to corresponded to a reduction in hospital length of stay, intensive care unit length of stay and cost of transfused blood products. (6)

2. Study objective 2.1 Primary Aim The aim of this study is to quantify the incidence of eTIC (defined as an elevated appt) and hyperfibrinolysis (defined as Ly30>7) in early trauma patients. To identify patients at risk of eTIC and hyperfibrinolysis, we will conduct a systematic search for trauma patients with an ISS>16 in whom a thrombelastogram (TEG) was obtained in the emergency department (ED)

The primary values of interest are:

* Initial activated partial thrombin time (appt)
* INR
* TEG (R time, MA, Lyseindex 30)

2.2 Secondary objectives

* Correlation of standard laboratory abnormalities (defined as an elevated appt) and TEG findings
* Correlation of eTIC and mortality
* Correlation of eTIC and blood product use in the first 24h

ELIGIBILITY:
Inclusion Criteria:

* Age < 18 years
* Sever trauma (ISS>16)
* Coagulation parameters (PT, aPTT, INR, fibrinogen, TEG) available within the first hour of admission

Exclusion Criteria:

* Patients with known pre-existing coagulopathies
* Patients on anticoagulant therapy prior to trauma
* Incomplete or missing coagulation data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with severe trauma (ISS>16)
Sampling Method: Non-Probability Sample
Enrollment: 263 (Actual)
Dates: Start 2025-05-25 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
incidence of eTIC | 1 hour after admission
  defined by increased appt/INR

SECONDARY OUTCOMES:
incidence of hyperfibrinolysis | 1 hour after admission
  defined as Ly30>7
Correlation of standard laboratory abnormalities and TEG findings | 1 hour after admission
  R and appt/INR MA and appt/INR K and appt/INR
Correlation of eTIC and mortality | 30 days
  eTIC defined by an increase of appt/INR

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Undecided